CLINICAL TRIAL: NCT02138019
Title: The Application of Fibrin Glue (Tissucol Duo Quick) in External Eye Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200910010M
Record Dates: First submitted 2011-07-01; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Corneal Ulcers; Cataract; Pterygium; Retinal Detachment
Keywords: corneal ulcers; conjunctival closure in strabismus surgery; surgery for retinal detachment; cataract surgery; mucous membrane grafting
MeSH Terms: conditions — Corneal Ulcer; Cataract; Pterygium; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fibrin glue (Experimental): In ophthalmic field, the use of organic glues has provided good results for the repair of leaking blebs and perforated corneal ulcers, conjunctival closure in strabismus surgery, surgery for retinal detachment, cataract surgery, trabeculectomy, and mucous membrane grafting to repair lesions of the conjunctival fornix. In this study, the investigators try to evaluate the effect of Fibrin Glue assisted external eye surgery.
  Interventions: Procedure: Fibrin Glue assisted external eye surgery; Device: Fibrin glue

INTERVENTIONS:
Procedure: Fibrin Glue assisted external eye surgery
Device: Fibrin glue

SUMMARY:
The fibrin sealants are prepared from fibrinogen, thrombin, and sometimes factor XIII that have been purified from human plasma. Tissucol Duo Quick (Baxter, Vienna, Austria) is a kind of fibrin sealants with popular use. It is a 2-component tissue adhesive that resembles natural fibrin formation. This glue has 2 components: fibrinogen (mixed with factor XIII and aprotinin) and thrombin-CaCl2 solution. When equal amounts of the 2 components are mixed, the monomers aggregate by cross-linking, resulting in a fibrin clot. It forms a elastic, whitish substance and provides strong adhesion to the tissue. Therefore, it is a good agent to seal small wounds or to replace the use of suture.

DETAILED DESCRIPTION:
Biologic adhesives have been used in medicine for many years. It has been applied to numerous surgical fields. As for the ophthalmic field, The use of organic glues has provided good results for the repair of leaking blebs and perforated corneal ulcers, conjunctival closure in strabismus surgery, surgery for retinal detachment, cataract surgery, trabeculectomy, and mucous membrane grafting to repair lesions of the conjunctival fornix. The fibrin sealants are prepared from fibrinogen, thrombin, and sometimes factor XIII that have been purified from human plasma. Tissucol Duo Quick (Baxter, Vienna, Austria)is a kind of fibrin sealants with popular use. It is a 2-component tissue adhesive that resembles natural fibrin formation. This glue has 2 components: fibrinogen (mixed with factor XIII and aprotinin) and thrombin-Calcium Chloride solution. When equal amounts of the 2 components are mixed, the monomers aggregate by cross-linking, resulting in a fibrin clot. It forms a elastic, whitish substance and provides strong adhesion to the tissue. Therefore, it is a good agent to seal small wounds or to replace the use of suture.

Pterygium is a triangular-shaped growth of abnormal conjunctival tissue that extends horizontally from the bulbar conjunctiva, across the limbus, and onto the cornea. Surgical removal is still the treatment of choice. Over the years, various treatment strategies such as simple excision with or without adjunctive measures (eg, postoperative [beta]-irradiation, intraoperative, and/or postoperative mitomycin C) and various techniques of conjunctival grafting have been tried to decrease recurrence after surgery. Conjunctival autograft and amniotic membrane transplantation are commonly used methods. However, they are time-consuming techniques because the graft must be fixed, usually by sutures. Tissue adhesives provide alternative ways for attaching conjunctival grafts and may shorten operating time, diminish postoperative discomfort, and remove suture-related complications. Using tissue adhesive instead of sutures results in shorter operation time. It has been reported by several studies. Furthermore, it seems also contributed to lower recurrence rate. National Taiwan University Hospital (NTUH), as one of the largest tertiary medical centers in Taiwan, is now in charge of a big part of difficult cases of ocular surface, including the refractory pterygium. With the previous experiences reported, the investigators are competent for this meaningful program to evaluate the effect and benefit of fibrin adhesives in external eye disease.

ELIGIBILITY:
Inclusion Criteria:

* It has been applied to numerous surgical fields.
* As for the ophthalmic field, The use of organic glues has provided good results for the repair of leaking blebs and perforated corneal ulcers, conjunctival closure in strabismus surgery, surgery for retinal detachment, cataract surgery,trabeculectomy,and mucous membrane grafting to repair lesions of the conjunctival fornix.

Exclusion Criteria:

* age: under 12 years and above 85 years
* cognitive impairment
* rejection from patients
* over size corneal ulcer (over 3mm)

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
pterygium recurrence | 12 months
  The grading system of postoperative recurrence of pterygium is as the follows: grade 1 with normal appearance of the operated site; grade 2 with the presence of fine episcleral vessels extending to the limbus, but no fibrous tissue; grade 3 with fibrovascular tissue in the excised area, reaching to the limbus but not invading the cornea; grade 4 with a true corneal recurrence, with fibrovascular tissue invading the cornea and across the limbus.

SECONDARY OUTCOMES:
Caruncular Morphology in Nasal Pterygia | 12 months
  A grading scale of 1 to 4 for the caruncle morphological characteristics was designed. Grade 1 with a normal appearance; grade 2 with synechia of conjunctival wound edge to the amniotic membrane covered area without change of caruncle location; grade 3 with thickened conjunctival wound edge without change of caruncular morphology; grade 4 with synechia of conjunctival wound edge to the amniotic membrane covered area with anterior advancement of caruncle location less than 3mm; grade 5 with synechia of conjunctival wound edge to the amniotic membrane covered area with anterior advancement of caruncle location more than 3mm.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD,PhD, Study Chair — NTUH
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan, Taiwan